CLINICAL TRIAL: NCT06400823
Title: Multimodal Platform Combining VR and TENS for Stroke Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute Mihajlo Pupin (Other)
Collaborators: ETH Zurich (Switzerland) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VRTENSSTROKE
Record Dates: First submitted 2024-04-19; First posted 2024-05-06 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-05

CONDITIONS: Stroke
Keywords: Virtual Reality; TENS; Stoke; Task-oriented rehabilitation; Multimodal intervention
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: The study has a parallel design, with two different groups.
  1. TENS+VR group
  2. Conventional therapy group
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VR+TENS (Experimental): Patients will undergo goal-oriented movements for upper-limb rehabilitation in a VR scenario. While performing the movement, patients will receive synchronous electrical stimulation targeting the medial nerve. The provided sensation will stimulate the interaction with elements in the virtual world.
  The intervention phase will last 3 weeks. Patients will undergo a minimum of three sessions per week (of around 60'). During each of these sessions, the first 10' will be employed for the calibration of the Transcutaneous Electrical Nerve Stimulation (TENS). In the remaining part of the session, subjects will perform some of the VR-based task-oriented games targeting different components.
  Interventions: Other: VR+TENS
- Conventional rehabilitation (Active Comparator): Patients in the control group will perform physical conventional rehabilitation provided by the rehabilitation clinic.
  The total amount of therapy will be the same as that of the VR+TENS group. The exercises will target the same components of the VR+TENS arm.
  Interventions: Other: Conventional rehabilitation

INTERVENTIONS:
Other: VR+TENS — During the invention, patients will be in VR scenarios and play task-oriented games, interacting with elements that appear in the virtual world, to improve mobility and functional independence of the upper limbs.
  The task-oriented games will target different components depending on the disability of the patient.
  Arms: VR+TENS
Other: Conventional rehabilitation — Patients will perform conventional upper-limb stroke rehabilitation. The movement performed will be comparable with the movement performed in the VR+TENS group
  Arms: Conventional rehabilitation

SUMMARY:
Stroke is a disabling medical condition annually affecting up to 15 million people worldwide. It leads to upper-limb impairments encompassing motor and sensory deficits together with cognitive self-body and space misrepresentation, overall limiting the functional independence of 70% of stroke survivors. On the motor side, stroke could account for hemiparesis (weakness or paralysis affecting the side contralateral to the brain lesion), muscle weakness, spasticity, loss of coordination, and others. On the sensory side, especially in the first stages after the stroke occurs, stroke could account for sensory loss, with the patient not being able to perceive what he's touching with the impaired arm.On a cognitive level, it has been shown that chronic stroke patients have distorted body representation and space representation. They perceive their impaired arm as shorter and the impaired hand as larger.

Despite initial evidence of the crucial role of sensory-motor integration toward a restored body representation to promote effective rehabilitation, conventional approaches suffer from the bias of prioritizing motor recovery, while disregarding stroke-induced sensory and body representation deficits.

In this view, the creation of a virtual reality (VR) scenario in which the person is fully immersed, could potentially play a significant role in improving stroke patients' rehabilitation.

Taking this into consideration, this project aims to assess whether a multimodal platform combining VR with TENS inducing full-body illusion toward a virtual avatar could positively impact motor performances, sensory assessments, and self-body and space representation of stroke patients.

More into detail, the intervention will consist of the patient performing some task-oriented movement within the virtual reality and congruently tactile receiving feedback through transcutaneous electrical nerve stimulation. The subject will receive clear instruction within the virtual reality scenario to perform specific actions toward a final goal. These actions will be designed to make the subject repeat some crucial movements in their rehabilitation process. Depending on the motor impairment of the patient, the investigators will adapt the characteristics and the difficulty of the task accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or haemorrhagic stroke patient
* At least 3 months after the stroke incident
* 10 <= FMUE <= 60 (motor function)

Exclusion Criteria:

* Prior neurological or psychiatric disorders
* Severe cognitive impairment (MoCA score <10)
* Epilepsy
* Pacemakers or other electronic implants
* Unable to give an informed consent form

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Changes in sensorimotor impairments | day 0 (before the first rehabilitation session, T0); 1.5 week (after six rehabilitation sessions, T1); 3 weeks (one day after the last rehabilitation session, T2); 5 weeks (2 weeks after the last rehabilitation session,T3)
  To assess the sensorimotor impairment in individuals who have had a stroke the investigators will use Fugl-Meyer for upper extremity (FMUE). FMUE assesses reflex activity, movement control, muscle strength, and sensory performances. It comprises items scored on a scale of 0 to 2, where 0 = cannot perform, 1 = performs partially and 2 = performs fully.
Changes in functional performances | day 0 (before the first rehabilitation session, T0); 1.5 week (after six rehabilitation sessions, T1); 3 weeks (one day after the last rehabilitation session, T2); 5 weeks (2 weeks after the last rehabilitation session,T3)
  To assess functional performance of the upper extremity through observational means the investigators will use the Action Research Arm Test (ARAT). The ARAT is a 19-item measure divided into 4 sub-tests (grasp, grip, pinch, and gross arm movement). The total score goes from 0 to 57. Performance on each item is rated on a 4-point ordinal scale ranging from: 3) Performs test normally 2) Completes test, but takes abnormally long or has great difficulty 1) Performs test partially 0) Can perform no part of test.
Changes in body-representation metrics | day 0 (before the first rehabilitation session, T0); 1.5 week (after six rehabilitation sessions, T1); 3 weeks (one day after the last rehabilitation session, T2); 5 weeks (2 weeks after the last rehabilitation session,T3)
  To measure the body representation of the subjects the investigators will use body-landmark metrics. In VR, the subject is asked to locate the position of specific body landmarks (e.g. elbow, inner wrist, outer wrist, index, ring) while a black panel is on top of his/her arm. The investigators will then compare the real and perceived dimensions of patients' arms and hands

SECONDARY OUTCOMES:
Changes in degree of assistance required by an individual | day 0 (before the first rehabilitation session, T0); 1.5 week (after six rehabilitation sessions, T1); 3 weeks (one day after the last rehabilitation session, T2); 5 weeks (2 weeks after the last rehabilitation session,T3)
  To assess the degree of assistance required by an individual on ten mobility and self-care the investigators will use the Barthel Index. The score goes from 0 to 100. It consists of an ordinal scale which measures a person's ability to complete activities of daily living (ADL).
Changes in peripersonal space | day 0 (before the first rehabilitation session, T0); 1.5 week (after six rehabilitation sessions, T1); 3 weeks (one day after the last rehabilitation session, T2); 5 weeks (2 weeks after the last rehabilitation session,T3)
  To measure the peri-personal space of stroke patients (the space in which multisensory integration is enhanced). Test Performance: In VR, the subject is sitting on a table and sees balls approaching him. He/she's asked to press a controller whenever he/she feels electrical stimulation.
Changes of spasticity indexes for shoulder, elbow and wrist | day 0 (before the first rehabilitation session, T0); 1.5 week (after six rehabilitation sessions, T1); 3 weeks (one day after the last rehabilitation session, T2); 5 weeks (2 weeks after the last rehabilitation session,T3)
  The investigators will use Ashworth Scale to test resistance to passive movement about a joint with varying degrees of velocity. This test is performed by extending the patients limb first from a position of maximal possible flexion to maximal possible extension (the point at which the first soft resistance is met).
Changes in pain perception | Every day, from day 1 to day 14; 5 weeks (2 weeks after the last rehabilitation session,T3)
  To quantify the experience of pain. This will be evaluated with Visual Analogue Scale. The score goes from 0 to 10.
Changes in neuropathic pain perception | day 0 (before the first rehabilitation session, T0); 1.5 week (after six rehabilitation sessions, T1); 3 weeks (one day after the last rehabilitation session, T2); 5 weeks (2 weeks after the last rehabilitation session,T3)
  To quantify the experience of pain. This will be evaluated with Neuropathic Pain Symptom Inventory (The score goes from 0 to 100)
Treatment Satisfaction Measure | 3 weeks (one day after the last rehabilitation session, T2)
  The subject marks on the treatment satisfaction on a Likert-scale.
Changes in tactile acuity | day 0 (before the first rehabilitation session, T0); 1.5 week (after six rehabilitation sessions, T1); 3 weeks (one day after the last rehabilitation session, T2); 5 weeks (2 weeks after the last rehabilitation session,T3)
  To measure the tactile acuity of patients we will use the Two-Point discrimination test. While blindfolded, the patient is repetitively touched with either one or two pins (fixed distance) and he asked to tell how many pins he/she feels.
Changes in upper-limb mobility (velocity) | Every day, from day 1 to day 14
  To assess changes in velocity the investigators will measure kinematic velocity of the patients while performing rehabilitation tasks.
Changes in upper-limb mobility (smoothness) | Every day, from day 1 to day 14
  To assess changes in smoothness the investigators will measure kinematic smoothness of the patients while performing rehabilitation tasks.
Changes in upper-limb mobility (efficiency) | Every day, from day 1 to day 14
  To assess changes in efficiency the investigators will measure the amount and rate of task-oriented movements of the patients.
Changes in upper-limb mobility (precision) | Every day, from day 1 to day 14
  To assess changes in precision the investigators will measure the spatial precision (error with respect to a predefined correct movement) during the task-oriented movements of the patient.

OTHER OUTCOMES:
Changes in cognitive abilities | day 0 (before the first rehabilitation session, T0); 1.5 week (after six rehabilitation sessions, T1); 3 weeks (one day after the last rehabilitation session, T2); 5 weeks (2 weeks after the last rehabilitation session,T3)
  To screen cognitive abilities and to detect mild cognitive dysfunction the investigators will use Montreal Cognitive Assessment (MoCA). The MoCA test is a one-page, 30-point test (score from 0 to 30) that can be administered in 10 minutes, assessing short-term memory recall, executive functions, concentration, attention, working memory and language.
Changes in neurophysiological correlates of Heart Rate | Every day, from day 1 to day 14
  Measure neurophysiological correlates of Heart Rate of the intervention. The subject will wear wrist wearable while performing the rehabilitation exercises.
Changes in neurophysiological correlates of Skin Conductance | Every day, from day 1 to day 14
  Measure neurophysiological correlates of Skin Conductance of the intervention. The subject will wear wrist wearable while performing the rehabilitation exercises.
Changes in brain connectivity | day 0 (before the first rehabilitation session, T0); 3 weeks (one day after the last rehabilitation session, T2)
  The patients will perform Functional Magnetic Resonance Imaging fMRI. Patients will perform baseline sessions of fMRI (patients not performing any task in the fMRI scanner).The outcome measures will be indexes of connectivity (graph analysis) in the somatosensory cortex.

CONTACTS AND LOCATIONS:
Overall Officials: Stanisa Raspopovic, PhD, Principal Investigator — Mihajlo Pupin Institute
Locations (1):
- Clinic for rehabilitation dr Miroslav Zotovic, Belgrade, Serbia

REFERENCES:
- [Background] Edwards LL, King EM, Buetefisch CM, Borich MR. Putting the "Sensory" Into Sensorimotor Control: The Role of Sensorimotor Integration in Goal-Directed Hand Movements After Stroke. Front Integr Neurosci. 2019 May 22;13:16. doi: 10.3389/fnint.2019.00016. eCollection 2019. PMID 31191265
- [Background] Bassolino M, Franza M, Guanziroli E, Sorrentino G, Canzoneri E, Colombo M, Crema A, Bertoni T, Mastria G, Vissani M, Sokolov AA, Micera S, Molteni F, Blanke O, Serino A. Body and peripersonal space representations in chronic stroke patients with upper limb motor deficits. Brain Commun. 2022 Aug 5;4(4):fcac179. doi: 10.1093/braincomms/fcac179. eCollection 2022. PMID 35950092
- [Background] Doyle S, Bennett S, Fasoli SE, McKenna KT. Interventions for sensory impairment in the upper limb after stroke. Cochrane Database Syst Rev. 2010 Jun 16;2010(6):CD006331. doi: 10.1002/14651858.CD006331.pub2. PMID 20556766
- [Background] Ingram LA, Butler AA, Brodie MA, Lord SR, Gandevia SC. Quantifying upper limb motor impairment in chronic stroke: a physiological profiling approach. J Appl Physiol (1985). 2021 Sep 1;131(3):949-965. doi: 10.1152/japplphysiol.00078.2021. Epub 2021 Jul 15. PMID 34264125
- [Background] Odermatt IA, Buetler KA, Wenk N, Ozen O, Penalver-Andres J, Nef T, Mast FW, Marchal-Crespo L. Congruency of Information Rather Than Body Ownership Enhances Motor Performance in Highly Embodied Virtual Reality. Front Neurosci. 2021 Jul 2;15:678909. doi: 10.3389/fnins.2021.678909. eCollection 2021. PMID 34295219
- [Background] Gladstone DJ, Danells CJ, Black SE. The fugl-meyer assessment of motor recovery after stroke: a critical review of its measurement properties. Neurorehabil Neural Repair. 2002 Sep;16(3):232-40. doi: 10.1177/154596802401105171. PMID 12234086
- [Background] Hsieh CL, Hsueh IP, Chiang FM, Lin PH. Inter-rater reliability and validity of the action research arm test in stroke patients. Age Ageing. 1998 Mar;27(2):107-13. doi: 10.1093/ageing/27.2.107. PMID 16296669
- [Background] Dworkin RH, Turk DC, Wyrwich KW, Beaton D, Cleeland CS, Farrar JT, Haythornthwaite JA, Jensen MP, Kerns RD, Ader DN, Brandenburg N, Burke LB, Cella D, Chandler J, Cowan P, Dimitrova R, Dionne R, Hertz S, Jadad AR, Katz NP, Kehlet H, Kramer LD, Manning DC, McCormick C, McDermott MP, McQuay HJ, Patel S, Porter L, Quessy S, Rappaport BA, Rauschkolb C, Revicki DA, Rothman M, Schmader KE, Stacey BR, Stauffer JW, von Stein T, White RE, Witter J, Zavisic S. Interpreting the clinical importance of treatment outcomes in chronic pain clinical trials: IMMPACT recommendations. J Pain. 2008 Feb;9(2):105-21. doi: 10.1016/j.jpain.2007.09.005. Epub 2007 Dec 11. PMID 18055266